CLINICAL TRIAL: NCT05661422
Title: Spectrographic and Acoustic Analysis of Lung Sounds Collected by RESP™ Biosensor to Support of Cardiorespiratory Therapeutic Decision Making in Monitored Hospitalized Pediatric Patients
Brief Title: Analysis of Lung Sounds Collected by RESP Biosensor to Support Decision Making in Monitored Hospitalized Pediatric Patients
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor Hold
Sponsor: Strados Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SL-MHUMC01
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Respiratory Diseases; Asthma; RSV Infection; COVID-19
MeSH Terms: conditions — Asthma; Respiratory Syncytial Virus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Participants
  Interventions: Device: RESP™ Biosensor

INTERVENTIONS:
Device: RESP™ Biosensor — The RESP Biosensor will be placed on the patient for periodic recording of auscultory sound.
  Other Names: RESP

SUMMARY:
This observational clinical trial is designed to confirm whether RESP™ Biosensor could be deployed to support clinical decision making in challenging pediatric cases, minimize clinician-to-clinician variability in lung sound interpretation, obviate the need to disrupt change of shift or chart rounds with physicians, and create a durable archive of the patient's lung sounds for longitudinal comparison within or across hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 4 and 17 with documented physician-diagnosed respiratory disease including infection such as RSV or COVID
2. Hospitalization projected for at least 24 hours after device placement
3. Patient and parent/guardian able and willing to provide informed consent/assent.

Exclusion Criteria:

1. Patient and parent/guardian unable or unwilling to provide informed consent
2. Patient expected to undergo prolonged invasive radiology procedure(s)
3. Plan for discharge within 24 hours
4. Patient expected to undergo major thoracic surgery
5. History of adverse reaction or allergy to TegaDerm ® or similar product

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric subjects who are admitted to the hospital with respiratory disease, including exacerbation of chronic respiratory disease and infection of RSV or COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Qualification and verification of lung sounds in pediatric population using RESP Biosensor | Periodic recording over 24 hours for inpatient stay

SECONDARY OUTCOMES:
Acceptability and utilization of RESP Biosensor in clinicians, healthcare staff and patient families | Periodic recording over 24 hours for inpatient stay
Limitations such as age in pediatric patients | Periodic recording over 24 hours for inpatient stay

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Health University Medical Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided